CLINICAL TRIAL: NCT02073097
Title: A Phase I/II Study of Carfilzomib in Combination With R-CHOP (CR-CHOP) for Patients With Diffuse Large B-cell Lymphoma
Brief Title: Carfilzomib, Rituximab, and Combination Chemotherapy in Treating Patients With Diffuse Large B-Cell Lymphoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CASE3413
Record Dates: First submitted 2014-02-25; First posted 2014-02-27 (Estimated); Results first posted 2024-05-29 (Actual); Last update posted 2024-05-29 (Actual); Status verified 2024-05

CONDITIONS: Contiguous Stage II Adult Diffuse Large Cell Lymphoma; Noncontiguous Stage II Adult Diffuse Large Cell Lymphoma; Stage I Adult Diffuse Large Cell Lymphoma; Stage III Adult Diffuse Large Cell Lymphoma; Stage IV Adult Diffuse Large Cell Lymphoma
MeSH Terms: conditions — Lymphoma, Large B-Cell, Diffuse | interventions — carfilzomib; Rituximab; Cyclophosphamide; Doxorubicin; Vincristine; Prednisone; pegfilgrastim; Granulocyte Colony-Stimulating Factor; Acyclovir

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- rituximab, combination chemotherapy, carfilzomib (Experimental): Participants receive (every 21 day cycle):
  * Rituximab IV over at least 90 minutes on day 2
  * Carfilzomib IV over 30 minutes on days 1, and 2
  * Cyclophosphamide IV over 30-60 minutes on day 3
  * Doxorubicin hydrochloride IV over 3-5 minutes on day 3
  * Vincristine sulfate IV over 1 minute on day 3
  * Prednisone PO on days 3-7 any time
  * Pegfilgrastim day 4
  * Acyclovir 2x per day from cycle 1, 6 months after completion of cycle 6
  Courses repeat every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Carfilzomib; Biological: Rituximab; Drug: Cyclophosphamide; Drug: Doxorubicin hydrochloride; Drug: Vincristine sulfate; Drug: Prednisone; Drug: Pegfilgrastim; Drug: Acyclovir

INTERVENTIONS:
Drug: Carfilzomib — Given IV, according to dose level. Cohorts begin with dose level (DL)1, escalated in standard 3+3 design to identify a recommended phase 2 dose DL (-2) 11 mg/m2 on day 1 and 2 every 21 days, cycles 1-6
  DL (-1) 15 mg/m2 on days 1 and 2 every 21 days, cycles 1-6
  DL (1) 20 mg/m2 days 1,2 every 21 days, cycles 1-6
  DL (2) 20 mg/m2 days 1,2 of cycle 1 followed by 27 mg/m2 days 1,2 every 21 days for cycles 2-6.
  DL (3) 20 mg/m2 days 1,2 of cycle 1 followed by 36 mg/m2 days 1,2 every 21 days for cycles 2-6.
  DL(4) 20 mg/m2 days 1,2 of cycle 1 followed by 45 mg/m2 days 1,2 every 21 days for cycles 2-6
  DL (5) 20 mg/m2 days 1,2 of cycle 1 followed by 56 mg/m2 days 1,2 every 21 days for cycles 2-6
  Other Names: Kyprolis; PR-171
Biological: Rituximab — Given IV (375mg/m^2)
  Other Names: IDEC-C2B8; IDEC-C2B8 monoclonal antibody; Mabthera; MOAB IDEC-C2B8; Rituxan
Drug: Cyclophosphamide — Given IV (750mg/m^2)
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: Doxorubicin hydrochloride — Given IV (50mg/m^2)
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: Vincristine sulfate — Given IV (1.4mg/m^2)
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: Prednisone — Given PO (100mg)
  Other Names: DeCortin; Deltra
Drug: Pegfilgrastim — 6 mg SC day 4 (every 21 days). Filgrastim 300 or 480 mcg IV/SC daily days 1-10 may be substituted if pegfilgrastim is not available. ONPROTM is also an acceptable method of administration.
  Other Names: Neulasta; Recombinant methionyl human granulocyte colony-stimulating factor (G-CSF)
Drug: Acyclovir — PO (400mg)
  Other Names: Zovirax

SUMMARY:
This phase I/II trial studies the side effects and best dose of carfilzomib when given together with rituximab and combination chemotherapy and to see how well they work in treating patients with diffuse large B-cell lymphoma. Carfilzomib may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as rituximab, can block cancer growth by finding cancer cells and helping kill them. Drugs used in chemotherapy work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. It is not known if carfilzomib in combination with R-CHOP is better or worse than R-CHOP alone in treating patients with diffuse large b-cell lymphoma.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the safety of carfilzomib in combination with rituximab-cyclophosphamide, doxorubicin hydrochloride, vincristine, and prednisone (R-CHOP) (CR-CHOP) in patients with newly diagnosed diffuse large B-cell lymphoma (DLBCL) and identify a recommended phase II dose (RP2D). (Phase I)

SECONDARY OBJECTIVES:

I. To determine if CR-CHOP improves the rates of 1-year progression free survival (PFS) and overall survival (OS) in non-germinal center (non-GC) DLBCL patients relative to historical controls treated with R-CHOP(Phase II) II. To determine response rates (complete and partial remission) in non-GC DLBCL patients treated with CR-CHOP and compare to historical controls treated with R-CHOP.

III. Because a proportion (~10%) of patients classified as non-GC by immunohistochemical (IHC) algorithms may not have the activated B-cells (ABC) subtyped of DLBCL, an exploratory secondary objective will compare the PFS, OS and response rates of the ABC subgroup of patients with DLBCL as determined by the Gene Expression Profiling with those of the overall group of non-GC DLBCL.

OUTLINE: This is a phase I, dose-escalation study of carfilzomib followed by a phase II study.

Patients receive rituximab intravenously (IV) over at least 90 minutes, cyclophosphamide IV over 30-60 minutes, doxorubicin hydrochloride IV over 3-5 minutes, vincristine sulfate IV over 1 minute on day 1, and prednisone orally (PO) on days 1-5. Patients also receive carfilzomib IV over 30 minutes on days 1, 2, 8 and 9. Courses repeat every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up at 30 days and at 6, 12, and 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed diffuse large B-cell lymphoma (DLBCL); patients with previously diagnosed indolent lymphoma (follicular lymphoma and marginal zone lymphoma but not small lymphocytic lymphoma) who have transformed to DLBCL are eligible only if they have not previously been treated for indolent lymphoma. For the Phase II study, patients must have non-GC DLBCL as determined by Hans Algorithm.
* Patients must have radiographically measurable disease
* Patients may have received brief (<15 days) treatment with glucocorticoids and/or 1 cycle of chemotherapy such as R-CHOP [or some component(s) thereof] for the diagnosis of B-cell lymphoma provided they had all necessary staging tests performed prior to R-CHOP including CT and/or PET/CT scans, echocardiogram and bone marrow biopsy. Treatment must occur within 60 days prior to enrollment.
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2; performance status of 3 will be accepted if impairment is caused by DLBCL complications and improvement is expected once therapy is initiated
* Hemoglobin ≥ 7.0 g/dl
* Absolute neutrophil count ≥ 1,500/mcL
* Platelet count ≥ 100,000/mcL
* Total bilirubin within normal institutional limits unless due to Gilbert's disease
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) ≤ 2.5 X institutional upper limit of normal
* Alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) ≤ 2.5 X institutional upper limit of normal
* Creatinine clearance ≥ 45 mL/min calculated by Cockcroft-Gault
* Adequate cardiac function left ventricular ejection fraction (LVEF) > 50% as assessed by echocardiogram or MUGA (Multi Gated Acquisition Scan)
* The effects of Carfilzomib on the developing human fetus are unknown. For this reason and because chemotherapeutic agents used in this study are known to be teratogenic, women of child-bearing potential and men must agree to use adequate contraception (double barrier method of birth control or abstinence) 2 weeks prior to initiation of treatment, for the duration of study participation and for 3 months after completing treatment. Should a woman become pregnant or suspect that she is pregnant while she or her partner is participating in this study, she should inform the treating physician immediately. Men must agree to refrain from sperm donation for at least 90 days after the last dose of carfilzomib.
* Subjects must have the ability to understand and the willingness to sign a written informed consent document
* International Prognostic Index must be documented:

  * ECOG performance status ≥ 2 (1 point)
  * Age ≥ 60 (1 point)
  * ≥ 2 extranodal sites (1 point)
  * Lactate dehydrogenase (LDH) > upper limit of normal (1 point)
  * Ann Arbor stage III or IV (1 point)

Exclusion Criteria:

* Patients who have not recovered from adverse events due to agents administered more than 4 weeks earlier
* Patients who are receiving any other investigational agents
* Known CNS involvement by lymphoma. Patients at high risk for secondary CNS involvement but without neurologic symptoms suspected to be due to lymphoma are allowed to be enrolled and receive intrathecal chemotherapy including but not limited to methotrexate, cytarabine and glucocorticoids. Patients who are enrolled and subsequently identified to have pathologic confirmation of CNS involvement by lymphoma may be continued on study at the discretion of the principal investigator.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to carfilzomib or other agents (R-CHOP) used in this study
* Active congestive heart failure (New York heart Association Class III or IV), symptomatic ischemia, or conduction abnormalities uncontrolled by conventional intervention or myocardial infarction within four months prior to enrollment
* Patients with uncontrolled intercurrent illness including, but not limited to ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study because Carfilzomib is a proteasome inhibitor with the potential for teratogenic or abortifacient effects. Because there is an unknown, but potential risk for adverse events in nursing infants secondary to treatment of the mother with Carfilzomib, breastfeeding should be discontinued if the mother is treated with Carfilzomib. These potential risks may also apply to other agents used in this study.
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with Carfilzomib. In addition, these patients are at increased risk of lethal infections when treated with marrow suppressive therapy. Appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated.
* Other malignancies within the past 3 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinomas of the skin, or low-risk prostate cancer after curative therapy, or low risk melanoma if treated with definitive therapy (such as excision) and expected to have a low likelihood of recurrence.
* Patients who have had major surgical procedures or significant traumatic injury within 28 days prior to study treatment
* Patients who are reported to be of direct Asian-Pacific (China, Japan, Taiwan, Singapore, Republic of Korea, and Thailand) ancestry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2015-01-28 (Actual); Primary Completion 2021-07-20 (Actual); Study Completion 2023-06-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Brian Hill, MD, PhD, Principal Investigator — Cleveland Clinic Taussig Cancer institute, Case Comprehensive Cancer Center
Locations (3):
- United States (3):
  - Roswell Park Comprehensive Cancer Center, Buffalo, New York
  - University Hospitals Cleveland Medical Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Cleveland Clinic Taussig Cancer Institute, Case Comprehensive Cancer Center, Cleveland, Ohio

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I CR-CHOP Level -2: Dose level -2:
  Carfilzomib: 11 mg/m^2 on day 1 and 2 every 21 days, cycles 1-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Level -1: Dose Level -1:
  Carfilzomib: 15 mg/m^2 on days 1 and 2 every 21 days, cycles 1-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Dose Level 1: Dose Level 1:
  Carfilzomib: 20 mg/m^2 days 1,2 every 21 days, cycles 1-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Dose Level 2: Dose Level 2:
  Carfilzomib: 20 mg/m^2 days 1,2 of cycle 1 followed by 27 mg/m^2 days 1,2 every 21 days for cycles 2-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Dose Level 3: Dose Level 3:
  Carfilzomib: 20 mg/m^2 days 1,2 of cycle 1 followed by 36 mg/m^2 days 1,2 every 21 days for cycles 2-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Dose Level 4: Dose Level 4:
  Carfilzomib: 20 mg/m^2 days 1,2 of cycle 1 followed by 45 mg/m^2 days 1,2 every 21 days for cycles 2-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
- Phase I CR-CHOP Dose Level 5; Phase II CR-CHOP Dose Level 5: Dose Level 5:
  Carfilzomib: 20 mg/m^2 days 1,2 of cycle 1 followed by 56 mg/m^2 days 1,2 every 21 days for cycles 2-6 CHOP: Standard dose on day 3 every 21 days Rituximab standard dose on Day 2
Period: Overall Study
Arm/Group | Phase I CR-CHOP Level -2 | Phase I CR-CHOP Level -1 | Phase I CR-CHOP Dose Level 1 | Phase I CR-CHOP Dose Level 2 | Phase I CR-CHOP Dose Level 3 | Phase I CR-CHOP Dose Level 4 | Phase I CR-CHOP Dose Level 5 | Phase II CR-CHOP Dose Level 5
Started | 0 | 0 | 9 | 3 | 3 | 3 | 6 | 24
Completed (Received at least 6 cycles of study drug.) | 0 | 0 | 9 | 3 | 3 | 3 | 6 | 18
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Physician Decision | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: All subjects who went on study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I CR-CHOP Level -2 | Phase I CR-CHOP Level -1 | Phase I CR-CHOP Dose Level 1 | Phase I CR-CHOP Dose Level 2 | Phase I CR-CHOP Dose Level 3 | Phase I CR-CHOP Dose Level 4 | Phase I CR-CHOP Dose Level 5 | Phase II CR-CHOP Dose Level 5 | Total
Number analyzed (Participants) | 0 | 0 | 9 | 3 | 3 | 3 | 6 | 24 | 48
Age, Customized [Count of Participants; unit: Participants]
  20-29 years old |  |  | 1 | 0 | 1 | 0 | 0 | 1 | 3
  30-39 years old |  |  | 1 | 0 | 0 | 0 | 1 | 2 | 4
  40-49 years old |  |  | 2 | 1 | 0 | 0 | 0 | 1 | 4
  50-59 years old |  |  | 2 | 1 | 1 | 1 | 2 | 5 | 12
  60-69 years old |  |  | 2 | 1 | 0 | 1 | 1 | 5 | 10
  70-79 years old |  |  | 1 | 0 | 1 | 1 | 2 | 10 | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female |  |  | 7 | 2 | 2 | 2 | 2 | 8 | 23
  Male |  |  | 2 | 1 | 1 | 1 | 4 | 16 | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Not Hispanic or Latino |  |  | 9 | 3 | 3 | 3 | 6 | 23 | 47
  Unknown or Not Reported |  |  | 0 | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White |  |  | 9 | 3 | 3 | 3 | 6 | 24 | 48
  More than one race |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported |  |  | 0 | 0 | 0 | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States |  |  | 9 | 3 | 3 | 3 | 6 | 24 | 48

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase II Dose (Phase I)
Description: Highest dose administered when no more than 1 out of 6 patients experience lose limiting toxicity below the maximally administered dose.
Time Frame: Through cycle 6 (each cycle is 21 days)
Population: The number of subjects that were on the phase I cohort.
Measure: Number; unit: mg/m^2
Arm/Group | Rituximab, Combination Chemotherapy, Carfilzomib
Number analyzed (Participants) | 24
mg/m^2
  Days 1, 2 of cycle 1 | 20
  Days 1, 2 every 21 days for cycles 2-6 | 56

2. Secondary Outcome: Progression Free Survival (Phase II)
Description: PFS will be estimated using a Kaplan-Meier curve. Progression-free Survival (PFS) is defined as the time from entry onto study until lymphoma progression or death from any cause. Participants was evaluated utilizing RECIST v1.0 criteria at baseline, 3 months after beginning treatment, end of treatment (6 cycles of therapy), and at 6 month, 12 month, and 24 month follow up visit. RECIST v1.0 criteria for Malignant Lymphoma use the following categories of response: Complete Response (CR), Partial Response (PR), Stable Disease (SD), Relapse and Progression (PD).
Time Frame: 31 months after treatment
Population: 24 participants were enrolled in Phase II.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Combination Chemotherapy, Carfilzomib
Number analyzed (Participants) | 24
percentage of participants | 79

3. Secondary Outcome: Overall Survival (Phase II)
Description: Overall survival will be estimated with a Kaplan-Meier curve. Overall survival is defined as the time from entry onto study until lymphoma progression or death from any cause.
Time Frame: 31 months after treatment
Population: 24 participants were enrolled to Phase II.
Measure: Number; unit: % of participants analyzed
Arm/Group | Rituximab, Combination Chemotherapy, Carfilzomib
Number analyzed (Participants) | 24
% of participants analyzed | 87

4. Secondary Outcome: Complete Response Rate (Phase II)
Description: The percentage of patients with a complete response as defined by a complete disappearance of all detectable clinical evidence of disease, and disease-related symptoms if present prior to therapy
Time Frame: 31 months after treatment
Population: 24 participants were enrolled to Phase II.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Combination Chemotherapy, Carfilzomib
Number analyzed (Participants) | 24
percentage of participants | 70

5. Secondary Outcome: Partial Response Rate (Phase II)
Description: The percentage of patients with a partial response as defined a >50% decrease in the sum of the product of the diameter of up to six of the largest nodes; no increase in the any node, liver, or spleen; no new sites of disease.
Time Frame: 31 months after treatment
Population: 24 participants were enrolled in Phase II.
Measure: Number; unit: percentage of participants
Arm/Group | Rituximab, Combination Chemotherapy, Carfilzomib
Number analyzed (Participants) | 24
percentage of participants | 19

ADVERSE EVENTS:
Time Frame: Adverse events were collected from time of participants on-study through follow-up (up to 31 months following treatment)
Description: All-cause mortality is zero for Phase I CR-CHOP Level -2 and Phase I CR-CHOP Level -1 because no participants were enrolled to these arms.
Arm/Group | Phase I CR-CHOP Level -2 | Phase I CR-CHOP Level -1 | Phase I CR-CHOP Dose Level 1 | Phase I CR-CHOP Dose Level 2 | Phase I CR-CHOP Dose Level 3 | Phase I CR-CHOP Dose Level 4 | Phase I CR-CHOP Dose Level 5 | Phase II CR-CHOP Dose Level 5
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 1/9 | 1/3 | 1/3 | 0/3 | 0/6 | 2/24
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 2/9 | 2/3 | 1/3 | 1/3 | 1/6 | 8/24
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 8/9 | 3/3 | 3/3 | 3/3 | 6/6 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I CR-CHOP Level -2 (N=0) | Phase I CR-CHOP Level -1 (N=0) | Phase I CR-CHOP Dose Level 1 (N=9) | Phase I CR-CHOP Dose Level 2 (N=3) | Phase I CR-CHOP Dose Level 3 (N=3) | Phase I CR-CHOP Dose Level 4 (N=3) | Phase I CR-CHOP Dose Level 5 (N=6) | Phase II CR-CHOP Dose Level 5 (N=24)
Anemia (Blood and lymphatic system disorders) | NA | NA | 1 | 0 | 0 | 1 | 0 | 1
Heart Failure (Cardiac disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 3
Diarrhea (Gastrointestinal disorders) | NA | NA | 0 | 1 | 0 | 1 | 0 | 1
Enterocolitis infectious (Infections and infestations) | NA | NA | 0 | 0 | 0 | 0 | 1 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | NA | NA | 0 | 0 | 0 | 0 | 1 | 2
Fever (General disorders) | NA | NA | 1 | 1 | 1 | 1 | 0 | 1
Gastric hemorrhage (Gastrointestinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 1 | 0
Hypotension (Vascular disorders) | NA | NA | 0 | 1 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | NA | NA | 0 | 1 | 0 | 0 | 0 | 1
Sinus tachycardia (Cardiac disorders) | NA | NA | 0 | 0 | 0 | 1 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | NA | NA | 0 | 1 | 0 | 0 | 0 | 1
Platelet count decreased (Investigations) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Infusion related reaction (General disorders) | NA | NA | 0 | 0 | 0 | 1 | 0 | 0
Lung Infection (Infections and infestations) | NA | NA | 0 | 1 | 0 | 0 | 0 | 1
Upper respiratory infection (Infections and infestations) | NA | NA | 1 | 0 | 0 | 0 | 0 | 0
Treatment related secondary malignancy (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | NA | NA | 1 | 0 | 0 | 0 | 0 | 0
Thromboembolic event (Vascular disorders) | NA | NA | 0 | 1 | 0 | 0 | 0 | 0
Atrial fibrillation (Cardiac disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Supraventricular tachycardia (Cardiac disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Infusion site extravasation (General disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Port containment (Infections and infestations) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Syncope (Nervous system disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Hematoma (Vascular disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Abdominal pain (Gastrointestinal disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Neutrophil count decreased (Investigations) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Hypercalcemia (Investigations) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
Chills (General disorders) | NA | NA | 0 | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase I CR-CHOP Level -2 (N=0) | Phase I CR-CHOP Level -1 (N=0) | Phase I CR-CHOP Dose Level 1 (N=9) | Phase I CR-CHOP Dose Level 2 (N=3) | Phase I CR-CHOP Dose Level 3 (N=3) | Phase I CR-CHOP Dose Level 4 (N=3) | Phase I CR-CHOP Dose Level 5 (N=6) | Phase II CR-CHOP Dose Level 5 (N=24)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Activated partial thromboplastin time prolonged (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Alanine aminotransferase increased (Investigations) | 0 | 0 | 2 | 1 | 1 | 0 | 1 | 3
Alkaline phosphatase increased (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 4 | 1 | 2 | 1 | 0 | 4
Anemia (Blood and lymphatic system disorders) | 0 | 0 | 3 | 2 | 2 | 1 | 2 | 7
Anorexia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 1
Aspartate aminotransferase increased (Investigations) | 0 | 0 | 3 | 2 | 1 | 0 | 1 | 3
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 2 | 1
Bloating (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Blurred vision (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 1 | 4
Breast pain (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Bruising (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Syncopal episode (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cerebrospinal fluid leakage (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Chest wall pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chills (General disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 2
Colitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 2 | 0 | 2 | 0 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 2 | 2 | 1 | 2 | 4
Diarrhea (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 0 | 2 | 2 | 8
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 1 | 1 | 1 | 0 | 4
Dry eye (Eye disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 4
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0 | 1 | 3 | 6
Impaired Balance (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Edema face (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Edema limbs (General disorders) | 0 | 0 | 0 | 0 | 2 | 2 | 1 | 4
Ejection fraction decreased (Investigations) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Eye Spasms (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 4 | 2 | 2 | 0 | 3 | 7
Fever (General disorders) | 0 | 0 | 0 | 2 | 1 | 1 | 0 | 3
Flank pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Flu like symptoms (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Gastroesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 2 | 2
Night Sweats (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Cold Sensitivity in Mouth (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Mental Fog (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 3
Headache (Nervous system disorders) | 0 | 0 | 2 | 1 | 1 | 0 | 0 | 3
Heart failure (Cardiac disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Hematoma (Vascular disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hematuria (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Hemoglobin increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hiccups (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Hypercalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Hyperglycemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 1
Hyperthyroidism (Endocrine disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 3
Hypocalcemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Hypokalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 6
Hypomagnesemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 1
Hyponatremia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2
Hypotension (Vascular disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 2
Yeast Infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Infusion related reaction (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2
Injection site reaction (General disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
INR increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 2 | 1 | 0 | 0 | 0 | 5
Elevated serum chloride (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Decreased Uric Acid (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritability (General disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Lymphocyte count decreased (Investigations) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 5
Elevated Glucose (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Middle ear inflammation (Ear and labyrinth disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Mitral valve disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Mucosal infection (Infections and infestations) | 0 | 0 | 1 | 0 | 1 | 1 | 0 | 2
Mucositis oral (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nail ridging (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 2 | 13
Neck edema (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0
Neutrophil count decreased (Investigations) | 0 | 0 | 5 | 0 | 0 | 1 | 2 | 2
Non-cardiac chest pain (General disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 1
Oral pain (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Pain (General disorders) | 0 | 0 | 3 | 0 | 2 | 0 | 0 | 5
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0
Palpitations (Cardiac disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Paresthesia (Nervous system disorders) | 0 | 0 | 3 | 0 | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1 | 0 | 2 | 0 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 0 | 0 | 5 | 0 | 0 | 2 | 3 | 9
Platelet count decreased (Investigations) | 0 | 0 | 3 | 0 | 1 | 1 | 2 | 5
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Presyncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Productive cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Rash acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 1
Urinary Hesitancy (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Chest congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Nasal Drainage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Sinus drainage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Intermittent Shortness of Breath (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Irritated Throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Scleral disorder (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Sinus tachycardia (Cardiac disorders) | 0 | 0 | 0 | 1 | 2 | 1 | 0 | 0
Sinusitis (Infections and infestations) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0
Skin Discoloration - RIght Leg (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Petechia - Abdomen from Lovenox (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin - Other - Peeling of skin of fingers (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin hyperpigmentation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Skin infection (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Insomnia (Social circumstances) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 1 | 2
Syncope (Nervous system disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1
Thromboembolic event (Vascular disorders) | 0 | 0 | 2 | 1 | 0 | 1 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Upper respiratory infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 0 | 0 | 1
Urinary frequency (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3
Urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 2
Voice alteration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 1 | 0 | 0 | 7
Weight gain (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
Weight loss (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
White blood cell decreased (Investigations) | 0 | 0 | 3 | 0 | 2 | 1 | 0 | 2
Hearing Impariment (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Malaise (General disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Flushing (Vascular disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Creatinine increased (Investigations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2
Renal and urinary disorders - Other (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Influenza (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Conjunctivitis (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Confusion (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Infections and infestations - Other (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
6 participants did not complete 6 cycles and were excluded from analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-09-01): https://cdn.clinicaltrials.gov/large-docs/97/NCT02073097/Prot_SAP_002.pdf
  • Informed Consent Form (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT02073097/ICF_001.pdf